CLINICAL TRIAL: NCT03700294
Title: A Phase 1, Open-Label, Dose-Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Antitumor Activity of ADCT-601 in Patients With Advanced Solid Tumors
Brief Title: Safety, Tolerability, Pharmacokinetics, and Antitumor Study of ADCT-601 to Treat Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Change in clinical plan and drug supply
Sponsor: ADC Therapeutics S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADCT-601-101
Record Dates: First submitted 2018-10-03; First posted 2018-10-09 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ADCT-601 (Experimental)
  Interventions: Drug: ADCT-601

INTERVENTIONS:
Drug: ADCT-601 — Intravenous (IV)

SUMMARY:
This study evaluates the safety, tolerance, pharmacokinetics (PK), and antitumor activity of ADCT-601 in patients with advanced solid tumors.

DETAILED DESCRIPTION:
This is a Phase 1 open-label, multicenter single-arm study with a dose-escalation phase (Part 1) followed by a dose-expansion phase (Part 2). The study will enroll approximately 75 patients. A standard 3+3 dose-escalation design will be used for Part 1 in order to determine the MTD and/or recommended dose for expansion (RDE).

Part 2 will consist of 3 cohorts from one or more selected tumor types. Each cohort will enroll 15 patients.

The study will include a Screening Period (of up to 28 days), a Treatment Period (cycles of 3-6 weeks), and a Follow-up Period (visits approximately every 12 weeks for up to 2 years after treatment discontinuation).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patient aged 18 years or older.
2. Pathologic diagnosis of one of the following solid tumor malignancies which is locally advanced or metastatic at screening:

   1. Breast cancer which is ER negative, partial response (PR) negative, and HER2 negative
   2. Colorectal cancer
   3. Esophageal cancer
   4. Gastric cancer
   5. Head and neck cancer (squamous cell carcinoma and nasopharyngeal carcinoma)
   6. Mesothelioma
   7. Non-small cell lung cancer
   8. Ovarian cancer
   9. Pancreatic cancer
   10. Soft Tissue Sarcomas
3. Patients with relapsed or refractory disease who have failed, or are intolerant to, any established therapy; or for whom no other treatment options are available, in the opinion of the Investigator.
4. Measurable disease per RECIST 1.1.
5. Patient must agree to biopsy of tumor for study biomarker testing.
6. Eastern Cooperative Oncology Group performance status, 0 to 1.
7. Adequate organ function as defined by screening laboratory values within the following parameters:

   1. Absolute neutrophil count (ANC) ≥ 1.5 × 103/µL (off growth factors at least 72 hours)
   2. Platelet count ≥100 x 103/µL without transfusion
   3. Alanine aminotransferase (ALT), aspartate aminotransferase (AST), and gamma glutamyl transferase (GGT) ≤ 2.5 × the upper limit of normal (ULN); ≤ 5 × ULN if there is liver involvement with tumor
   4. Total bilirubin ≤ 1.5 × ULN (patients with known Gilbert's syndrome may have a total bilirubin up to ≤ 3 × ULN)
   5. Blood creatinine ≤ 1.5 × ULN or calculated creatinine clearance ≥ 60 mL/min by the Cockcroft and Gault equation.
8. Negative beta-human chorionic gonadotropin (β-HCG) pregnancy test within 7 days prior to start of study drug (C1D1) for women of childbearing potential.
9. Women of childbearing potential must agree to use a highly effective method of contraception from the time of giving informed consent until at least 16 weeks after the last dose of ADCT-601. Men with female partners who are of childbearing potential must agree that they will use a highly effective method of contraception from the time of giving informed consent until at least 16 weeks after the patient receives his last dose of ADCT-601.

Exclusion Criteria:

1. Known history of ≥ Grade 3 hypersensitivity to a therapeutic antibody.
2. Active second primary malignancy other than nonmelanoma skin cancers, nonmetastatic prostate cancer, in situ cervical cancer, ductal or lobular carcinoma in situ of the breast, or other malignancy that the Sponsor's medical monitor and Investigator agree and document should not be exclusionary.
3. Active autoimmune disease, including motor neuropathy considered of autoimmune origin and other central nervous system (CNS) autoimmune disease. Patients with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll, provided the trigger can be avoided.
4. Known seropositive and requiring antiviral therapy for human immunodeficiency virus, hepatitis B virus, or hepatitis C virus.
5. History of Stevens-Johnson syndrome or toxic epidermal necrolysis.
6. Symptomatic CNS metastases or evidence of leptomeningeal disease (brain MRI or previously documented cerebrospinal fluid cytology).

   Previously treated asymptomatic CNS metastases are permitted provided that the last treatment (systemic anticancer therapy and/or local radiotherapy) was completed ≥ 8 weeks prior to Day 1 except usage of low dose of steroids on a taper (ie, up to 10 mg on Day 1 and consecutive days is permissible if being tapered down). Patients with discrete dural metastases are eligible.
7. Clinically significant third space fluid accumulation (ie, ascites requiring drainage or pleural effusion that is either requiring drainage or associated with shortness of breath).
8. Breastfeeding or pregnant.
9. Significant medical comorbidities, including but not limited to, uncontrolled hypertension (blood pressure [BP] ≥ 160/100 mmHg repeatedly), unstable angina, congestive heart failure (greater than New York Heart Association class II), electrocardiographic evidence of acute ischemia, coronary angioplasty or myocardial infarction within 6 months prior to screening, uncontrolled atrial or ventricular cardiac arrhythmia, poorly controlled diabetes, or severe chronic pulmonary disease.
10. Major surgery, radiotherapy, chemotherapy, or other antineoplastic therapy within 14 days prior to start of study drug (C1D1), except shorter if approved by the Sponsor.
11. Use of any other experimental medication within 14 days prior to start of study drug (C1D1).
12. Planned live vaccine administration after starting study drug (C1D1).
13. Failure to recover to Grade ≤1 (Common Terminology Criteria for Adverse Events [CTCAE] version 4.0) from acute non-hematologic toxicity (Grade ≤ 2 neuropathy or alopecia) due to previous therapy prior to screening.
14. Congenital long QT syndrome or a corrected QTcF interval of > 480 ms at screening (unless secondary to pacemaker or bundle branch block).
15. Any other significant medical illness, abnormality, or condition that would, in the Investigator's judgment, make the patient inappropriate for study participation or put the patient at risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-12-21 (Actual); Primary Completion 2019-12-11 (Actual); Study Completion 2019-12-11 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicity | First 21 to 42 - day cycle for each patient depending if patient is treated every 3, 4 or 6 weeks (dose escalation only)
  Frequency and severity of adverse events (AEs) and serious adverse events (SAEs)
Maximum Tolerated Dose | Treatment cycle is every 3-6 weeks. Patients followed every 12 weeks for up to 2 years after treatment
  Incidence of dose-limiting toxicities (DLTs) and frequency of dose interruptions and dose reductions

SECONDARY OUTCOMES:
Overall response rate (ORR) | Up to 2 Years
  According to the Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 defined as the proportion of patients with a best overall response (BOR) of complete response (CR) or partial response (PR).
Disease control rate (DCR) | Up to 2 years
  According to the RECIST 1.1 defined as the proportion of patients with a BOR of CR, PR, or SD.
Duration of response (DOR) | Up to 2 years
  Defined as the time from the documentation of first tumor response to disease progression or death.
Overall survival (OS) | Up to 2 years
  Defined as the time between the start of treatment and death from any cause.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Sarah Cannon Research Institute at HealthONE, Denver, Colorado
  - Florida Cancer Specialists, Sarasota, Florida
  - The Sarah Cannon Research Institute (Tennessee Oncology), Nashville, Tennessee
  - NEXT Oncology, San Antonio, Texas